CLINICAL TRIAL: NCT01701232
Title: A Multicenter Open-label Randomized Study of BCD-020 (Rituximab, CJSC BIOCAD, Russia) Efficacy and Safety in Comparison With MabThera (F. Hoffmann-La Roche Ltd., Switzerland) in Monotherapy of CD20-positive Indolent Non-Hodgkin's Lymphoma
Brief Title: Safety and Efficacy Study of BCD-020 in Therapy of Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIORIX (BCD-020-3)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Follicular Non-Hodgkin's Lymphoma; Nodal Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma
Keywords: lymphoma, non-Hodgkin's
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MabThera (Active Comparator): Reference rituximab at a dose of 375 mg/m2 intravenously once a week for four weeks (on days 1, 8, 15 and 22)
  Interventions: Biological: rituximab
- BCD-020 (Experimental): Proposed rituximab biosimilar at a dose of 375 mg/m2 intravenously once a week for four weeks (on days 1, 8, 15 and 22)
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — Patients will receive rituximab at a dose of 375 mg/m2 intravenously once a week for 4 weeks (on day 1,8,15,22)
  Other Names: Biological: BCD-020, MabThera

SUMMARY:
This international multi-center, randomized, controlled, open-label study investigated the pharmacokinetics, pharmacodynamics, efficacy and safety of BCD-020 (INN: rituximab, CJSC Biocad) versus MabThera® (INN: rituximab, F. Hoffmann La Roche, Ltd.) both administered as a monotherapy of patients with indolent non-Hodgkin's lymphoma.

Patients were randomized to receive 375 mg/m² BCD-020 as intravenous infusion once a week for 4 weeks or MabThera® at the same regimen.

ELIGIBILITY:
Inclusion Criteria:

* Having signed a written informed consent;
* Patients' age is 18 years or more;
* Diagnosis of CD20-positive indolent non-Hodgkin lymphoma of following morphological types:Follicular non-Hodgkin lymphoma stage II-IV according to Ann Arbor, grade I-II;Nodal marginal zone lymphoma stage II-IV according to Ann Arbor; Splenic marginal zone lymphoma.
* Life expectancy of not less than 3 months after the enrollment in the study;
* Morphological and immunohistochemical examination of the tumor (both lymph node biopsy and bone marrow biopsy) - within 3 months before the enrollment in the study ;
* Performance status ≤2 on the ECOG scale;
* Hemoglobin > 80 g/l; leukocyte count ≥ 3.0×109/l but less than 25×109/l, absolute neutrophil count ≥1.5×109/l, platelet count ≥100×109/l;
* Presence of at least one measurable lesion;
* Patient's ability in the investigator's opinion to comply with the protocol procedures;
* Willingness of patients with preserved reproductive function to use reliable contraception methods (at least two contraception methods in women, e.g., spermicide and condom).

Exclusion Criteria:

* Bulky disease - size of any single lesion more than 10 cm in the greatest diameter;
* Secondary transformation to high-grade lymphoma;
* Other types of non-Hodgkin lymphomas apart from follicular non-Hodgkin stage II-IV lymphoma according to Ann Arbor, grade 1,2; nodal marginal zone lymphoma stage II-IV according to Ann Arbor; splenic marginal zone lymphoma.
* Patients regularly taking corticosteroids during 1 month preceding the enrollment in the study;
* Occurrence of other (aside from NHL) diseases that can distort the assessment of the main disease symptoms expression; mask, enhance, modify the main disease symptoms or induce clinical and laboratory-instrumental symptoms similar to the non-Hodgkin lymphomas; Severe resistant hypertension; Decompensated forms of heart (NYHA class ХСН III, IV), liver and kidney disorders (creatinine level >133 µmol/l, AST, ALT, and bilirubin level 3 times exceeding the norm) except for the cases where the symptom is caused by lymphoma; Decompensated respiratory failure; Tumor infiltration of the lungs; Decompensated diabetes mellitus; Active autoimmune diseases; Ongoing infections requiring antimicrobial therapy.
* Usage of the drugs:

At any time prior to the enrollment into the study - interferon-based drugs or monoclonal antibodies for the treatment of NHL; Chemotherapy or radiotherapy was completed less than 21 day prior to the enrollment into the study; Vaccination within 1 week prior to the enrollment into the study;

* Presence of any psychiatric disorders including major depressive conditions and/or suicidal thoughts in anamnesis that in opinion of the investigator may put a patient at an excessive risk or influence the ability of patients to fulfill the study protocol;
* Myocardial infarction less than 1 month before the enrollment into the study;
* Severe CNS or PNS dysfunctions;
* Drug and alcohol addiction;
* Known HIV, HBV, HCV infection, syphilis;
* Known primary or secondary immunodeficiency;
* Primary CNS lymphoma or metastasis in the CNS;
* Known intolerance or allergy to mouse proteins or any components of the study drugs, and also to the premedication drugs;
* Pregnancy or lactation;
* Prior or concomitant malignances except for adequately treated basal cell carcinoma and in situ cervical cancer;
* Any restraints or impossibility to administer the study drug via an intravenous infusion;
* Major surgery within 1 week prior to the enrollment into the study;
* Simultaneous participation in any other clinical study or any preceding participation in other studies within 3 months prior to enrollment in this study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2011-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | day 50 (cycle 4)
  Estimation of the overall response rate in each treatment arm at the end of treatment
CD20-positive cells count | day 50
  Comparison of peripheral blood B-cell depletion and repletion after BCD-020 and MabThera intravenous administration

SECONDARY OUTCOMES:
Cmax | day 22
  Estimation of maximum rituximab serum concentrations after administration of BCD-020 to that obtained after administration of MabThera
AUC(0-168) | 168 hours
  Estimation of rituximab exposition after administration of BCD-020 to that obtained after administration of MabThera
Complete response rate | day 50
  Assessment of complete response rates of BCD-020 and MabThera given as a monotherapy at the end/completion of the treatment
Frequency of AEs/sAEs grade 3-4 (CTCAE v.4.03) | day 50
  Evaluation of the safety profiles of BCD-020 and MabThera
Levels of binding and neutralizing antibodies to rituximab | day 50
  Immunogenicity assessment of BCD-020 and MabThera
AUC(0-1176), AUC(0-inf) | day 50
  Estimation of rituximab serum concentrations after administration of BCD-020 to that obtained after administration of MabThera

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD,MD, Study Director — CJSC Biocad
Locations (62):
- Colombia (3):
  - Instituto Nacional de Cancerología, Bogotá
  - Fundación Reina Isabel, Cali
  - Hospital Pablo Tobon Uribe, Medellín
- India (19):
  - HCG Multi Specialty Hospitals, Ahmedabad
  - Department of Medical Oncology, Navneet Memorial Hospital, "Sushrusha", Ahmedabad
  - Sujan Surgicals, Amaravati
  - HCG Bangalore Institute of Oncology, Bangalore
  - Department of Medicine (Haemotology), St.John's Medical College Hospital, Bangalore
  - Narayana Hrudayalaya Hospitals, Bangalore
  - Srinivasam Cancer Care Hospital, Bangalore
  - All India Institute of medical Sciences (AIIMS), Bhubaneswar
  - Acharya Tulasi Regional Cancer Treatment and Research Centre, Bikaner
  - G.Kuppuswamy Naidu Memorial Hospital, Coimbatore
  - Medical Oncology Department, The Karnatak Cancer Therapy and Research Institute, Hubli
  - BIBI General hospital & cancer center, Hyderabad
  - Department of Medical Oncology, Basavatarakam Indo-American Cancer Hospital and Research Institute, Hyderabad
  - Omega Hospitals, Hyderabad
  - Nilratan Siracar Medical College & Hospital, Kolkata
  - King George Medical University, Lucknow
  - Department of Radiation Oncology, Meenakshi Mission Hospital & Research Centre, Madurai
  - Manas Super Speciality Hospital, Nashik
  - City Cancer Center, Vijayawada
- Russia (36):
  - Arkhangelsk District Clinical Oncology Dispensary, Arkhangelsk
  - City Hospital N8, Barnaul
  - Public health facility "Irkutsk Regional Oncology Center", Irkutsk
  - Ivanovo Regional Oncology Center, Ivanovo
  - State Health Care Institution "Republican Clinical Cancer Center," the Ministry of Health of the Udmurt Republic, Izhevsk
  - Public health facility "Kemerovo Regional Hospital", Kemerovo
  - Clinical Oncology Dispensary N1, Krasnodar
  - Public health facility "Kursk Regional Cancer Center," Health Committee of Kursk region, Kursk
  - Public health facility "Lipetsk Regional Oncology Center", Lipetsk
  - N.N. Burdenko General Military Clinical Hospital, Moscow
  - Russian Medical Academy of Post-Graduate Education, Ministry of Health and Social Development of the Russian Federation, Moscow
  - Research Center for Hematology MHSD RF, Moscow
  - Official body of the health of the city of Moscow "Moscow City Clinical Hospital named after S. P. Botkin", Moscow
  - Medical Radiological Research Center, Ministry of Health and Social Development of the Russian Federation, Obninsk
  - Regional government health care "Oryol Regional Hospital", Oryol
  - Perm Region Oncology Dispensary, Perm
  - V.A. Baranov Republican Hospital of Ministry of Health republic Karelia, Petrozavodsk
  - Pyatigorsk Oncology Center, Pyatigorsk
  - Russian Research Institute of Hematology and Transfusiology Federal State Institution of Federal Medical and Biological Agency, Saint Petersburg
  - St. Petersburg State Health Care Institution "Alexander City Hospital", Saint Petersburg
  - Saint Petersburg City Clinical Oncology Center, Saint Petersburg
  - Saint Petersburg Pavlov State Medical University, Saint Petersburg
  - V.A. Almazov Federal Center for Heart, Blood and Endocrinology, Ministry of Health and Social Development of the Russian Federation, Saint Petersburg
  - N.N.Petrov Oncology Research Center, Saint Petersburg
  - Russian scientific center of radiology and surgery technologies, Saint Petersburg
  - The federal government military educational institution of higher education, "Military Medical Academy named after SM Kirov's' Ministry of Defense", Saint Petersurg
  - Provincial health official body "Smolensk Regional Clinical Oncological Dispensary", Smolensk
  - Oncology Dispensary 2, Sochi
  - Tambov Regional Oncology Center, Tambov
  - Municipal Health "Clinical Hospital № 5" Togliatti, Tolyatti
  - Tula Regional Hospital, Tula
  - Public health care setting of the Tyumen region "Regional Oncology Center", Tyumen
  - State Health Care Institution Republican Clinical Hospital named after G. G. Kuvatova, Ufa
  - Republican Clinical Oncology Dispensary of Ministry of Health republic Bashkortostan, Ufa
  - Volgograd District Oncology Dispensary №1, Volgograd
  - Municipal Institution "Central City Hospital № 7", Yekaterinburg
- Medi-Clinic Vereeniging, Vereeniging, South Africa
- Ukraine (3):
  - Khmel'nyts'kyy Regional Hospital, Hematology Department, Khmelnytskyi
  - National Cancer Institute of Ukraine, Oncohematology Department, Kiev
  - State Institution "Institute of Blood Pathology and Transfusion Medicine AMS of Ukraine", Hematology Department, Lviv

IPD SHARING:
Plan to Share IPD: No